CLINICAL TRIAL: NCT06035302
Title: Madany Closure: A Novel Technique for Fascial Closure in Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ClinAmygate (Other)
Collaborators: Aswan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR00C1940
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cholecystolithiasis
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Madany closure (Experimental): the novel port site closure technique is to be done for this group
  Interventions: Procedure: Madany Closure
- Control (Active Comparator): external closure of the port site
  Interventions: Procedure: Standard closure

INTERVENTIONS:
Procedure: Madany Closure — Madany Closure is a new technique for the porte site closure
  Arms: Madany closure
Procedure: Standard closure — Standard closure technique of the port site from ecternal
  Arms: Control

SUMMARY:
this study aims to evaluate the effectiveness of the use of a basic laparoscopic instrument (Only needle holder) with a new technique for port site closure

ELIGIBILITY:
Inclusion Criteria:

* age . 18 years
* eligible for Laparoscopic cholecystectomy

Exclusion Criteria:

* refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
closure time | 1 day
  closure time in seconds
rate of closure failure | 1 day
  rate failure to close the port site

SECONDARY OUTCOMES:
incidence of port site infection | 1 month
  incidence of infection of the port site
incidence of port site hernia | 6 weeks
  incidence of hernia at the port site

CONTACTS AND LOCATIONS:
Overall Officials: Mohie El-Din M Madani, MD, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University Hospital, Aswān, Egypt